CLINICAL TRIAL: NCT00745836
Title: Effects of Atorvastatin on Adiponectin Levels and Insulin Sensitivity In Hypercholesterolemic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Model: Parallel | Purpose: Treatment
Other Study IDs: GMC-200508
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Hypercholesterolemia
Keywords: insulin sensitivity
MeSH Terms: conditions — Hypercholesterolemia; Insulin Resistance | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- atorvastatin 10 mg, 80 mg (Experimental)
  Interventions: Drug: statin

INTERVENTIONS:
Drug: statin

SUMMARY:
High dose atorvastatin may worsen insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* hypercholesterolemia

Exclusion Criteria:

* chronic renal disease

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Derived] Koh KK, Quon MJ, Han SH, Lee Y, Kim SJ, Shin EK. Atorvastatin causes insulin resistance and increases ambient glycemia in hypercholesterolemic patients. J Am Coll Cardiol. 2010 Mar 23;55(12):1209-1216. doi: 10.1016/j.jacc.2009.10.053. PMID 20298928